CLINICAL TRIAL: NCT00767299
Title: Effects of Arzoxifene on Bone Mineral Density in Korean Postmenopausal Women With Osteoporosis
Brief Title: A Study of Arzoxifene to Treat Korean Women With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12185; H4Z-MC-GJAV
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — LY 353381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: arzoxifene
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: arzoxifene — 20 mg, QD, PO,24 weeks
  Other Names: LY353381
  Arms: 1
Drug: Placebo — QD, PO, 24 weeks
  Arms: 2

SUMMARY:
The study is for Korean women who are postmenopausal and also suffer from osteoporosis.

The study will test if women who are given 20 mg of arzoxifene once a day for six months have a less severe level of osteoporosis than those women who do not take arzoxifene.

All patients will receive 500 mg of elemental calcium and 400 to 600 IU Vitamin D daily starting 4 weeks prior to study drug administration continuing through the 6 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Present with osteoporosis based on total hip, femoral neck or lumbar spine BMD T-score of less than or equal to -2.5 but must never have had any osteoporotic fragility fracture.
* Are ambulatory and are 60 to 85 years of age, inclusive. Aside from diagnosed osteoporosis (Inclusion Criterion [1]), all women must be free of severe or chronically disabling conditions, have a life expectancy of at least 5 years in the opinion of the investigator, be expected to remain ambulatory throughout the entire study, and be expected to return for follow-up visits.
* Had their last natural menstrual period at least 2 years before beginning the study.
* Are able to comprehend the requirements and procedures for the study and to provide informed consent before entering the study.
* Have at least two lumbar vertebrae (L1 to L4) that are evaluable via dual energy X-ray absorptiometry (DXA) and lateral thoracic and lumbar spine x-ray films that can be adequately evaluated for existing vertebral fractures at screening.
* Have centrally read total hip, femoral neck or lumbar spine T-score less than or equal to -2.5

Exclusion Criteria:

* Have known current metabolic bone disorders other than low bone mass, such as hyperparathyroidism, renal osteodystrophy, or osteomalacia.
* Have known, suspected, or history of carcinoma of the breast or estrogen-dependent neoplasia (e.g., endometrial or uterine carcinoma), except for hysterectomized patients with a history of carcinoma in situ of the uterus. For other cancers, be disease free and in remission from all other cancers for 5 or more years, except for excised superficial lesions, such as basal cell carcinoma or squamous cell carcinoma of the skin.
* Have demonstrated or suspected allergy to raloxifene or arzoxifene
* Have unexplained or abnormal vaginal bleeding within 6 months prior to Visit 1 or between Visit 1 and Visit 2.
* Are experiencing clinically severe postmenopausal symptoms that may require estrogen-replacement therapy.
* Have a history of or suggestion on ultrasound or pelvic examination of a pre-existing gynecologic abnormality that would require further gynecologic treatment (e.g., ovarian cysts, large fibroids, undiagnosed adnexal masses) or of baseline endometrial thickness of >5 mm.
* Have Papanicolaou's tests showing malignant or premalignant findings.
* Have active or any past history of thromboembolic events
* Have active or any past history of atrial fibrillation.
* Have a history of cerebrovascular accident or documented transient ischemic attack at any time in the past.
* Have acute or chronic liver disease defined as alanine aminotransaminase (ALT) >100 U/L, gamma-glutamyl transferase (GGT) >400 U/L, or late stage cirrhosis without transaminase elevations.
* Have impaired kidney function (serum creatinine >177 micromol/L or >2.0 mg/dL).
* Have vitamin D deficiency prior to enrollment (Visit 2; 25-hydroxyvitamin D less than10 ng/mL or less than 24.9 nmol/L).
* Have any known, severe, or untreated malabsorption syndromes.
* Have endocrine disorders requiring pharmacologic therapy except for type II diabetes and hypothyroidism. Patients on a stable dose of thyroid replacement therapy during the 6 months preceding randomization (Visit 2) who are clinically euthyroid in the opinion of the investigator may enroll in the trial.
* Consume an excess of alcohol or abuse drugs
* Represent an unacceptable medical or psychiatric risk for treatment with an investigational drug
* Have active or any history of seizure disorder.

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Lumbar spine bone mineral density (BMD), by dual energy X-ray absorptiometry (DXA) analyses | 6 months

SECONDARY OUTCOMES:
Incidence of spontaneous vaginal bleeding. | 6 months
Total hip BMD | 6 months
Biochemical marker of bone metabolism (serum CTX and PINP) | 3 and to 6 months
Overall safety of arzoxifene administration in Korean postmenopausal women | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul